CLINICAL TRIAL: NCT04788381
Title: The Effects of Preoperative Bevacizumab on Perioperative Complications in Patients With Tumor Undergoing Unexpected Operation
Brief Title: The Effects of Preoperative Bevacizumab on Perioperative Complications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Suzhanzhang, Director of Cancer Institute of Zhejiang University, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: RWS-CRC-LC-S
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer; Lung Cancer; Operation Wound; Infection; Bevacizumab
Keywords: bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Surgical Wound Infection | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with CRC or lung cancer was performed unexpected operation: This is an observational study; thus, no intervention or treatment is required by the protocol. During the study, enrolled patients may be eligibled if bevacizumab was discontinued within 6 weeks prior to unexpected operation.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Enrolled patients may be eligibled if bevacizumab was discontinued within 6 weeks prior to unexpected operation.
  Other Names: Avastin

SUMMARY:
This is a nationwide multicenter,retrospective,observational real-world study.

1. To assess the risk of perioperative complications in patients with tumor who received bevacizumab prior to unexpected operation.
2. To assess the correlation of the interval time between the last dose of bevacizumab and operation and occurrence of perioperative complications.
3. To explore the risk factors of perioperative comlications in patients with tumor received bevacizumab prior to unexpected operation.

DETAILED DESCRIPTION:
Avastin (bevacizumab) is a recombinant humanized monoclonal IgG1 antibody that binds to and inhibits the biologic activity of human vascular endothelial growth factor(VEGF) in in vitro and in vivo assay systems. Bevacizumab was first granted marketing approval in the United States on 26 February 2004 (international birth date) in combination with IV 5-fluorouracil(5-FU) based chemotherapy for the first-line treatment of patients with metastatic carcinoma of the colon or rectum (CRC). At present, bevacizumab is widely used in the treatment of solid tumors such as lung cancer ,colorectal cancer and so on. It has been reported in the literature that bevacizumab may adversely affect wound healing. To prevent postoperative complications, some guidelines state that the interval time between last dose of bevacizumab and operations should be at least 6 weeks, but the optimal time to discontinue bevacizumab before surgery has not been confirmed. This project aims to evaluate the risk of perioperative complications in cancer patients with a history of bevacizumab use within 6 weeks prior to unexpected operation.

This is a nationwide multicenter,retrospective,observational real-world study.The study will collect the medical records and prognosis in 30 days following surgery of patients with colorectal cancer and lung cancer who underwent unexpected operation within 6 weeks (including 6 weeks) of bevacizumab discontinuation from 01 Jan 2010 to 31 Dec 2019.All enrolled subjects aged 18-90 years old; Complete clinical data related to important indicators, including preoperative baseline data, surgical information and perioperative prognosis information. The patients who used anti-angiogenic agents other than bevacizumab within 6 weeks prior to surgery would be excluded.

Primary Evaluation Measures: To assess the risk of perioperative complications in patients with tumor who received bevacizumab prior to unexpected operation:to calculate the total incidence of perioperative complications in patients undergoing unexpected surgery after discontinuation of bevacizumab, including wound healing complications, non-wound-related infections, postoperative bleeding, thrombosis, gastrointestinal perforation, anastomotic leakage, secondary surgery, death and other perioperative adverse events;to calculate the incidence of each perioperative complication in patients undergoing unexpected operation after bevacizumab discontinuation.

SAS9.4 statistical analysis software will be used for analysis. Measurement indicators will be statistically described using number of cases, mean, median, standard deviation, minimum and maximum; categorical indicators will be statistically described using frequency and percentage. Unless otherwise specified, all statistical tests will adopt the two-sided test with α = 0.05, and the corresponding OR value and two-sided 95% confidence interval will be provided if applicable.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with colorectal cancer and lung cancer who underwent unexpected operation from 01 Jan 2010 to 31 Dec 2019, and received bevacizumab within 6 weeks (including 6 weeks) before operation;
* 2.Patients aged 18-90 years old;
* 3.Complete clinical data related to important indicators, including preoperative baseline data, surgical information and perioperative prognosis information.

Exclusion Criteria:

* Patients who used anti-angiogenic agents other than bevacizumab within 6 weeks prior to unexcepted operation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with colorectal canceror lung cancer who underwent unexpected operation within 6 weeks (including 6 weeks) of bevacizumab discontinuation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
To assess the risk of perioperative complications in patients with tumor who received bevacizumab prior to unexpected operation. | 30 days after operation
  To calculate the total incidence of perioperative complications in patients undergoing unexpected surgery after discontinuation of bevacizumab, including wound healing complications, non-wound-related infections, postoperative bleeding, thrombosis, gastrointestinal perforation, anastomotic leakage, secondary surgery, death and other perioperative adverse events;To calculate the incidence of each perioperative complication in patients undergoing unexpected operation after bevacizumab discontinuation.

SECONDARY OUTCOMES:
To assess the correlation of the interval time between the last dose of bevacizumab and operation and occurrence of perioperative complications. | 30 days after operation
  According to the interval between the last dose of preoperative bevacizumab and surgery, the patients were divided into three groups: within 2 weeks (including 2 weeks), 2 weeks to 4 weeks (including 4 weeks), and 4 weeks to 6 weeks (including 6 weeks). If the number of patients actually enrolled in each group was too small to support subsequent analysis, the grouping was adjusted according to the interval between the last dose of preoperative bevacizumab and surgery, such as two groups: within 4 weeks, 4 weeks to 6 weeks, or the possibility of other grouping, depending on the actual enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Su Zhan Zhang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China